CLINICAL TRIAL: NCT01558752
Title: A Randomized Clinical Trial of a Modular Cementless Acetabular Metal on Poly Component Versus a Monoblock Cementless Titanium Shell With Ceramic on Ceramic Bearing and CORAIL Stem: A Bone Mineral Density Study
Brief Title: A Clinical Trial of a Metal on Poly Component Versus CORAIL Stem: A Bone Mineral Density Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2010913-01H
Record Dates: First submitted 2012-03-16; First posted 2012-03-20 (Estimated); Results first posted 2020-12-19 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-11

CONDITIONS: Total Hip Arthroplasty
Keywords: Total Hip Replacement; Bone Mineral Density; Stem; Dual-energy x-ray absorptiometry; DXA-RFA; Corail; Tri-Lock
MeSH Terms: interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Titanium Shell with CORAIL stem (Experimental): Patients in Group 1 will receive a total hip replacement with titanium shell and CORAIL stem.
  Interventions: Device: Total hip replacement with titanium shell and CORAIL stem
- Modular Titanium Femoral Stem (Tri-Lock) (Active Comparator): Patients in Group 2 will receive a total hip replacement with Modular Titanium Femoral Stem (Tri-lock).
  Interventions: Device: Total hip replacement with Modular Titanium Femoral Stem

INTERVENTIONS:
Device: Total hip replacement with titanium shell and CORAIL stem — Patients that are randomized into Group 1 will receive a total hip replacement with the following components: CORAIL (impaction broach) titanium stem and a monoblock cup with ceramic on ceramic bearing (DELTA motion).
  Arms: Titanium Shell with CORAIL stem
Device: Total hip replacement with Modular Titanium Femoral Stem — Patients that are randomized into Group 2 will receive a total hip replacement with the following components: the Trilock-Pinnacle system (titanium stem and titanium cup with polyethylene insert).
  Arms: Modular Titanium Femoral Stem (Tri-Lock)

SUMMARY:
The main goal is to prospectively evaluate bone mineral density adjacent to the femoral component and femoral bone remodeling of two different designs: CORAIL impaction broach titanium stem compared to a modular titanium femoral stem (Tri-lock). Patients will be randomized to one of the two treatment groups prior to surgery. Each patient will be evaluated at their regularly scheduled 10-14 days, 3, 6, 12 and 24 month visits following surgery. Patients will be asked to have bilateral DEXA bone mineral density tests (10-14 days post-surgery, and 6, 12 and 24 months post-operatively). Urine and serum samples (measures of bone turnover) will be collected at 3, 6 and 12 months post-operatively after an overnight fast. Patient reported questionnaires will be completed preoperatively and at the 3, 6, 12, and 24 month visits.

DETAILED DESCRIPTION:
The main goal is to prospectively evaluate bone mineral density adjacent to the femoral component and femoral bone remodeling of two different designs: CORAIL impaction broach titanium stem compared to a modular titanium femoral stem (Tri-lock). The investigators expect the CORAIL femoral stem group to show significantly less bone loss on the femoral side as compared to the Tri-lock group. The primary outcome is percent change in bone mineral density (BMD) (g/cm2) from baseline (10-14 days post-op) to the two year post-operative interval, as measured radiographically in zones 1 and 7.

Patients will be randomized to one of the two treatment groups prior to surgery. Each patient will be evaluated at their regularly scheduled 10-14 days, 3, 6, 12 and 24 month visits following surgery.

Bilateral DXA bone mineral density tests will be performed at 10-14 days following surgery (baseline assessment) and at 6, 12, and 24 months post-operatively.

Urine and serum samples (measures of bone turnover) will be collected at 3, 6 and 12 months post-operatively after an overnight fast.

The Harris Hip Score will be completed at each post-operative visit except the immediate (10-14 days), when risk of dislocation precludes a determination of range of motion. At the 3, 6, 12 and 24 month post-operative visits, the patient will complete the SF-36 Item Health Survey, WOMAC and UCLA activity scale.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are undergoing primary hip surgery for osteo/degenerative arthritis (does not include traumatic arthritis, congenital hip dysplasia, or avascular necrosis).
* Patients who are skeletally mature, as determined by Risser sign or at least 18 years of age
* Patients under 75 years of age
* Patients for whom there is a reasonable expectation that they will be available for each examination scheduled over a two year post-operative follow-up period.

Exclusion Criteria:

* Patients with previous fusions, acute femoral neck fractures and above knee amputations.
* Patients with evidence of active local infection
* Patients with neurologic or musculoskeletal disease that may adversely affect gait or weight-bearing.
* Patients who have previously undergone an ipsilateral hemi resurfacing, total resurfacing, total bipolar, unipolar or total hip replacement device, or any prior hip surgery or retained internal fixation.
* Patients who are anticipated to require contralateral hip surgery in the next year
* Patients with known disorders of bone metabolism, systemic inflammatory disorders, and use of drug medications, including oral steroids, HRT, Tamoxifen, calcium, or vitamin D in the past year, and any past bisphosphonate therapy.
* Patients with a Body Mass Index (BMI) > 35
* Patients with neuropathic joints
* Patients with severe documented psychiatric disease
* Patients requiring structural bone grafts
* Patients with an ipsilateral girdlestone
* Patients with sickle cell disease
* Patients with major acetabular bone stock deficiency

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2010-04 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2020-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul E Beaulé, MD, FRCSC, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital - General Campus, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Slullitel PA, Mahatma MM, Farzi M, Grammatopoulos G, Wilkinson JM, Beaule PE. Influence of Femoral Component Design on Proximal Femoral Bone Mass After Total Hip Replacement: A Randomized Controlled Trial. J Bone Joint Surg Am. 2021 Jan 6;103(1):74-83. doi: 10.2106/JBJS.20.00351. PMID 33079901
- [Derived] Fischman D, Mahatma MM, Slullitel P, Farzi M, Grammatopoulos G, Poitras S, Wilkinson JM, Beaule PE. Does a Monoblock Acetabular Component With a Ceramic Liner Cause More Pelvic Bone Loss Than a Conventional Modular Cementless Acetabular Component? A 2-Year Randomized Clinical Trial. J Arthroplasty. 2022 Jan;37(1):75-82. doi: 10.1016/j.arth.2021.08.033. Epub 2021 Sep 4. PMID 34649747

RESULTS

PARTICIPANT FLOW:
Groups:
- Corail: Patients in Group 1 will receive a total hip replacement with titanium shell and CORAIL stem.
  Total hip replacement with titanium shell and CORAIL stem: Patients that are randomized into Group 1 will receive a total hip replacement with the following components: CORAIL (impaction broach) titanium stem and a monoblock cup with ceramic on ceramic bearing (DELTA motion).
- Tri-Lock: Patients in Group 2 will receive a total hip replacement with Modular Titanium Femoral Stem (Tri-lock).
  Total hip replacement with Modular Titanium Femoral Stem: Patients that are randomized into Group 2 will receive a total hip replacement with the following components: the Trilock-Pinnacle system (titanium stem and titanium cup with polyethylene insert).
Period: Overall Study
Arm/Group | Corail | Tri-Lock
Started | 42 | 46
Completed | 40 | 46
Not Completed | 2 | 0
Not completed — Physician Decision | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Corail | Tri-Lock | Total
Number analyzed (Participants) | 40 | 46 | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (10.2) | 60.4 (10.1) | 59.4 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 24 | 47
  Male | 17 | 22 | 39
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 40 | 46 | 86
American Society of Anesthesiologists (ASA) Grade [Count of Participants; unit: Participants] — The ASA grade is a physical status classification system that is used for assessing the fitness and co-morbidities of patients before surgery. Patients are categorized between grades 1-6, with a lower grade indicative of better health and less co-morbidities.
  Participants
    Grade 1 | 3 | 1 | 4
    Grade 2 | 31 | 28 | 59
    Grade 3 | 6 | 17 | 23

OUTCOME MEASURES:

1. Primary Outcome: Change in Bone Mineral Density
Description: To prospectively evaluate bone mineral density adjacent to the femoral component and femoral bone remodeling for the 2 groups. Bone mineral density was assessed using high-sensitivity dual x-ray absorptiometry region-free analysis (DXA-RFA). Mean number of pixels with change with significant BMD decrease.
Time Frame: 2 Years Post-operative
Measure: Mean (Standard Deviation); unit: number of pixels with change
Arm/Group | Corail | Tri-Lock
Number analyzed (Participants) | 40 | 46
number of pixels with change | 1072 (50) | 1295 (73)

2. Secondary Outcome: Comparison of Bone Turnover Markers Between Groups
Description: Biochemical markers of bone turnover will be assessed from morning-fasting serum samples and compared from baseline to 2-years post-operative.
Time Frame: 2 Years post-operative
Reporting Status: Not Posted

3. Secondary Outcome: Implant Migration
Description: Stem and cup migration will be assessed using radiographic images at baseline and 2-years post-operative.
Time Frame: 2 years post-operative
Reporting Status: Not Posted

4. Secondary Outcome: Change in Modified Harris Hip Score
Description: The change from baseline to 2-years post-operative on the Modified Harris Hip Score (mHHS). The mHHS assesses a patient's functional outcome and pain. The maximum score is 100 and the lowest is 0. A higher score is indicative of better outcomes and lower pain levels.
Time Frame: 2 Years post-operative
Reporting Status: Not Posted

5. Secondary Outcome: Change in SF-36 Score
Description: The change from baseline to 2-years post-operative on the SF-36 score: a quality of-life measure. The score consists of 36 questions separated into 8 concepts. These outcomes will be grouped as physical component summary and mental component summary. The norm data is 0-100. The health related quality of life is increases as the scores are increased. The average score is 50.
Time Frame: 2 Years post-operative
Reporting Status: Not Posted

6. Secondary Outcome: Change in WOMAC Questionnaire
Description: The change from baseline to 2-years post-operative on the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC). The WOMAC score consists of 24 items, separated into 3 subscales. Each question is scored on a scale of 0 to 4, with a possible score range of 0-20 for pain, 0-8 for stiffness, and 0-68 for physical function. The scores of each subscale are summed to give a total score. Higher scores are indicative of worse pain, stiffness and functional limitations.
Time Frame: 2 Years post-operative
Reporting Status: Not Posted

7. Secondary Outcome: Change in UCLA Activity Scale
Description: The change from baseline to 2-years post-operative on the UCLA Activity score. The UCLA activity scale is a 10 point scale evaluating a patients activity level. The possible score range is from 0-10. A low value is indicative of sedentary or inactivity, whereas a high score is indicative of high levels of activity.
Time Frame: 2 Years post-operatively
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data was collected at each standard of care clinical visit (10-14 days post-op, 3-, 6-, 12- and 24-months post-operative).
Arm/Group | Corail | Tri-Lock
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/46
Serious Adverse Events (participants affected / at risk) | 1/40 | 1/46
Other Adverse Events (participants affected / at risk) | 4/40 | 7/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Corail (N=40) | Tri-Lock (N=46)
Superficial wound infection (Infections and infestations) | 1 (1) | 0 (0) — Superficial wound infection 1 month post-op requiring irrigation and debridement (I&D) surgery.
Aseptic Loosening (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Aseptic loosening is considered a relatively common complication of hip joint replacements. The patient generally experiences a great deal of pain and requires revision surgery.
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Corail (N=40) | Tri-Lock (N=46)
Thigh pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5) — Participants that reported greater than normal pain levels in the thigh area.
Intra-operative Calcar Fracture (Metabolism and nutrition disorders) | 3 (3) | 1 (1) — The incidence of intraoperative calcar fractures, a known complication of total hip arthroplasty (THA).
Femoral nerve palsy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Femoral nerve dysfunction is a loss of movement or sensation in parts of the legs due to damage to the femoral nerve and is a complication that occurs during surgery.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-02-07): https://cdn.clinicaltrials.gov/large-docs/52/NCT01558752/Prot_SAP_000.pdf